CLINICAL TRIAL: NCT00325325
Title: A Pilot Study to Investigate Pharmacokinetic Characteristics of Everolimus in Patients Treated With Tacrolimus-Based Immunosuppression in De Novo Kidney Transplantation
Brief Title: Pharmacokinetic Study on the Combination of Everolimus-Tacrolimus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Novartis (Industry); Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVEROTAC
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-05

CONDITIONS: Kidney Diseases
Keywords: Kidney Transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — Everolimus; Tacrolimus

INTERVENTIONS:
Drug: everolimus and tacrolimus

SUMMARY:
The purpose of this study is to address the pharmacokinetic (PK) profiles of everolimus and tacrolimus in combination in de novo kidney transplant recipients, comparing 1.5 and 3 mg per day of everolimus in fixed doses. For comparison purposes, pharmacokinetic profiles will be performed at first dose (abbreviated), 4th day, 14th day, and 42nd day post-transplantation.

DETAILED DESCRIPTION:
To address the pharmacokinetic profiles of everolimus and tacrolimus in combination in de novo kidney transplant recipients, comparing 1.5 and 3 mg per day of everolimus in fixed doses. For comparison purposes, pharmacokinetic profiles will be performed at first dose (abbreviated), 4th day, 14th day, and 42nd day post-transplantation. Patients will receive triple therapy steroids, tacrolimus and everolimus. Tacrolimus will be administered at a dose of 0.15 mg/kg/day to achieve 10-15 ng/ml 14 days, and 5-10 thereafter. During the first 6 weeks (the PK study period) everolimus will be assigned to fixed dose of 0.75 or 1.5 mg bid. After day 42, everolimus will be adjusted for 3-8 ng/ml and tacrolimus minimized to optimize graft function. Efficacy and safety parameters at 6 months post-transplantation will be secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients aged 18-65 years old with a presumed immediately functioning graft

Exclusion Criteria:

* Non-functioning kidneys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2007-06

PRIMARY OUTCOMES:
12-hour PK profiles of everolimus and tacrolimus on day 14 post-transplantation with everolimus 1.5 mg versus 3 mg per day

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pascual, MD, Study Chair — Hospital Universitario Ramon y Cajal; Gorka G Erauzquin, MD, Principal Investigator — Hospital de Cruces, Bilbao; José M Morales, MD, Principal Investigator — Hospital 12 de Octubre, Madrid; Luis Pallardó, MD, Principal Investigator — Hospital Dr Peset, Valencia; Ricardo Lauzurica, MD, Principal Investigator — Hospital Germans, Trias i Puyol, Badalona; Domingo del Castillo, MD, Principal Investigator — Hospital Reina Sofía, Córdoba; Josep M Grinyó, MD, Principal Investigator — Hospital de Bellvitge, Barcelona
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain